CLINICAL TRIAL: NCT04691934
Title: Our Anesthesia Experiences in COVID-19 Positive Patients Undergoing Cesarean Section: A Retrospective Single-center Cohort Study
Brief Title: Obstetric Anesthesia Experiences in COVID-19 Positive Patients
Status: Completed | Type: Observational
Sponsor: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Derya Karasu, MD, Assoc Prof., Turkiye Yuksek Ihtisas Education and Research Hospital
Other Study IDs: U1111-1263-2201
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Obstetric Anesthesia
Keywords: COVID-19; Anesthesia; Cesarean Section; Pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Anesthesia management — Patients who underwent cesarean section and had positive PCR nasopharyngeal swabs for COVID-19 were included in the study. Patients who tested negative and were clinically suspicious were excluded from the study. PCR test was not performed on all elective and emergency pregnant women to be taken for cesarean section in our hospital. It was only applied to patients with symptoms or patients who were suspected. All patient demographics and information about anesthesia were analyzed retrospectively from the patient files.

SUMMARY:
At the end of 2019, a new coronavirus named COVID-19 (SARS-CoV-2), one of the lower respiratory tract samples was detected in China. The World Health Organization (WHO) declared it a global epidemic on March 11, 2020, due to the emergence of COVID-19 cases in 113 countries other than China, where the first epidemic occurred, and the spread and severity of the virus. Pregnancy increases susceptibility to respiratory complications of viral diseases.

This study aimed to retrospectively evaluate the demographic data of COVID-19 patients undergoing cesarean section, our anesthesia practices, complications, and condition of neonates, and to summarize up-to-date information on COVID-19 in obstetric anesthesia.

DETAILED DESCRIPTION:
Our study was a single-center, retrospective, and observational trial and carried out with the principles of the Declaration of Helsinki. All patient demographics and information about anesthesia were analyzed retrospectively from the patient files.

All patients were operated in negative pressure operating theatres reserved for them. The whole team was equipped with Level 3 personal protective equipment (PPE) (liquid-proof apron, N-95 mask, goggles, visor, overshoes). Anesthesia was administered by 2 healthcare professionals from the anesthesia team, including an experienced anesthesiologist and an assistant anesthesia technician. A third person was kept ready outside to help in case of need.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent cesarean section
* Patients who had positive PCR nasopharyngeal swabs for COVID-19

Exclusion Criteria:

* Patients who tested negative and were clinically suspicious

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients who underwent cesarean section were included in the study
Study Population: Patients who underwent cesarean section and had positive PCR nasopharyngeal swabs for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
obstetric anesthesia practices | until 30 minutes after arrival in the operating room
  the type of anesthesia was investigated

SECONDARY OUTCOMES:
anesthesia complications | up to 1 hour after anesthesia
  hypotension, nausea, vomiting, allergies

CONTACTS AND LOCATIONS:
Overall Officials: Derya Karasu, Principal Investigator — BursaYuksek Ihtisas Training and Research Hospital
Locations (1):
- University of Health Sciences Turkey, Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Yıldırım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided